CLINICAL TRIAL: NCT01918475
Title: Analgesic Effect of Oxytocin Receptor Modulation in Healthy Volunteers
Brief Title: Analgesic Effect of Oxytocin Receptor Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 140/12; 2013DR1021 (Other: Swissmedic)
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Pain; Hyperalgesia; Central Sensitization
Keywords: randomized controlled trial; placebo controlled trial; cross over trial
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbetocin first (Active Comparator): Subjects receive carbetocin 0.1 mg intravenously in the first session and placebo (NaCl 0.9%) in the second session
  Interventions: Drug: Carbetocin; Drug: Placebo
- Placebo first (Active Comparator): Subjects receive placebo (NaCl 0.9%) intravenously in the first session and carbetocin 0.1 mg in the second session
  Interventions: Drug: Carbetocin; Drug: Placebo

INTERVENTIONS:
Drug: Carbetocin — Carbetocin 0.1 mg single dose is intravenously administered
Drug: Placebo — 1ml of NaCl 0.9% is administered intravenously

SUMMARY:
Carbetocin is a synthetic analogue of the hormone Oxytocin and is routinely used in obstetric anesthesiology to control uterine bleeding after cesarean section. As an incidental finding, women who received carbetocin had less pain after cesarean section than women who had received Oxytocin. Carbetocin may therefore have an analgesic effect.

The present study examines this analgesic effect using different sensory tests, e.g. pressure, heat, cold and electrical pain before and after administration of carbetocin in healthy male volunteers. Any changes in these sensory tests might be indicative of an analgesic property of carbetocin.

DETAILED DESCRIPTION:
Background

Chronic pain is still a largely unresolved issue, causing suffering, disability and high social costs. The search for novel pharmacological targets is therefore a priority. A recent study on postpartal bleeding came to the accidental finding of a possible analgesic action of the oxytocin agonists carbetocin.

Oxytocin is a well known nonapeptide synthesized in the hypothalamus, acting as neurohormone during parturition and the milk ejection reflex. Animal studies have found that descending pathways for oxytocin synthetizing neurons project to the lamina I-II of the spinal cord, where they activate a subpopulation of glutamatergic and GABAergic interneurons. In addition to GABAergic hyperpolarisation, models of oxytocin selectively blocking A-delta and C-fibers have been published. Intrathecal administration of oxytocin prevents long-term potentiation in the dorsal horn, which is thought to be an important mechanism of enhanced central pain processing.

Antagonism to GABAergic and glycinergic neurotransmission mimics many symptoms of inflammatory and neuropathic pain. A loss of synaptic inhibition in the dorsal horn occurs in animal models of experimental pain.

Inhibitory synaptic transmission in the spinal cord dorsal horn use GABA and glycine as their principal fast neurotransmitters. Both of them open the Cl- -channels, which induce postsynaptic hyperpolarisation and impairs the propagation of excitatory potentials on dendrites of neurons. Immunofluorescence studies have revealed abundant glycinergic innervations in the dorsal horn. According to this model, inhibitory GABAergic and glycinergic interneurons in the superficial spinal dorsal horn are key components in the control of pain transmission from the periphery to the brain. The model states that a non-painful stimulation is felt as non painful as long as the synaptic GABAergic and glycinergic inhibition remains intact. A human study on GABAergic modulation of pain by benzodiazepines has been recently performed by our group and was suggestive for an analgesic action. However, these drugs cause sedation and addiction, which strongly limit their clinical usefulness. A pharmacological GABA modulation via the oxytocin receptor may be an attractive alternative, since oxytocin agonists are devoid of these side effects.

Quantitative sensory tests (QST) are used to explore the central processing of painful stimuli in healthy volunteers and patients. They are based on a multimodal and multi-tissue approach, combining different pain modalities applied to different tissues in order to gather sufficient and differentiated information about the human nociceptive system under normal and pathological conditions. QST will be our tool to characterize analgesic efficacy of carbetocin.

Objective

We will test the hypothesis that carbetocin produces analgesia in healthy volunteers, as assessed by multimodal experimental pain testing.

Methods

Intradermal capsaicin injection in the volar forearm is used to create experimental pain an hyperalgesia. The area of hyperalgesia to pinprick and brush allodynia is quantified, and pressure, heat, cold and electrical pain thresholds as well as nociceptive withdrawal reflex thresholds are assessed 30 minutes after capsaicin injection (baseline assessments). Carbetocin 0.1 mg is injected intravenously and the above measurements repeated after 10, 60 and 120 minutes. Blood samples are taken in order to investigate plasma carbetocin levels at 10, 60 and 120 minutes and genetic variants of the oxytocin receptor gene.

ELIGIBILITY:
Inclusion Criteria:

* male
* pain-free
* written informed consent

Exclusion Criteria

* chronic pain
* acute pain at time of testing
* sign or suspicion of neurological dysfunction at the tested sites
* intake of opioids
* intake of benzodiazepines
* intake of antidepressants
* intake of anticonvulsants
* intake of any analgesic drug 48h prior to test
* known allergy to carbetocin
* allergy to capsaicin
* cardiovascular disease
* asthma bronchiale
* migraine
* epilepsy
* history of liver disease
* history of renal disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in intramuscular electrical pain threshold compared to baseline | 10, 60 and 120 minutes after carbeoticin administration

SECONDARY OUTCOMES:
Capsaicin-induced area of hyperalgesia and allodynia | 10, 60 and 120 minutes after carbeoticin administration
Nociceptive withdrawal reflex thresholds of the foot | 10, 60 and 120 minutes after carbeoticin administration
Single cutaneous electrical pain thresholds | 10, 60 and 120 minutes after carbeoticin administration
Repeated cutaneous electrical pain thresholds | 10, 60 and 120 minutes after carbeoticin administration
Single intramuscular electrical pain threshold | 10, 60 and 120 minutes after carbeoticin administration
Heat pain detection threshold | 10, 60 and 120 minutes after carbeoticin administration
Heat pain tolerance threshold | 10, 60 and 120 minutes after carbetocin administration

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, M.D., Ph.D., Study Chair — University Department of Anesthesiology and Pain Therapy, Inselspital Bern, Switzerland
Locations (1):
- University Department of Anesthesiology and Pain Therapy, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] De Bonis M, Torricelli M, Leoni L, Berti P, Ciani V, Puzzutiello R, Severi FM, Petraglia F. Carbetocin versus oxytocin after caesarean section: similar efficacy but reduced pain perception in women with high risk of postpartum haemorrhage. J Matern Fetal Neonatal Med. 2012 Jun;25(6):732-5. doi: 10.3109/14767058.2011.587920. Epub 2011 Jul 15. PMID 21761999
- [Background] Rousselot P, Papadopoulos G, Merighi A, Poulain DA, Theodosis DT. Oxytocinergic innervation of the rat spinal cord. An electron microscopic study. Brain Res. 1990 Oct 8;529(1-2):178-84. doi: 10.1016/0006-8993(90)90825-v. PMID 2282492
- [Background] Breton JD, Veinante P, Uhl-Bronner S, Vergnano AM, Freund-Mercier MJ, Schlichter R, Poisbeau P. Oxytocin-induced antinociception in the spinal cord is mediated by a subpopulation of glutamatergic neurons in lamina I-II which amplify GABAergic inhibition. Mol Pain. 2008 May 29;4:19. doi: 10.1186/1744-8069-4-19. PMID 18510735